CLINICAL TRIAL: NCT01984424
Title: A Double-blind, Randomized, Multicenter Study to Evaluate the Safety and Efficacy of Evolocumab, Compared With Ezetimibe, in Hypercholesterolemic Subjects Unable to Tolerate an Effective Dose of a HMG-CoA Reductase Inhibitor Due to Muscle Related Side Effects
Brief Title: Goal Achievement After Utilizing an Anti-PCSK9 Antibody in Statin Intolerant Subjects-3
Acronym: GAUSS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120332; 2013-000935-29 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Hyperlipidemia
Keywords: High Cholesterol, Treatment for high cholesterol, Lowering cholesterol, Lowering high cholesterol, Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe; evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A: Atorvastatin 20 mg => Placebo (Other): Participants received atorvastatin 20 mg orally for 10 weeks (period 1) followed by placebo orally for 10 weeks (period 2), separated by a 2-week washout period.
  Interventions: Drug: Atorvastatin; Drug: Placebo to Atorvastatin
- Part A: Placebo => Atorvastatin 20 mg (Other): Participants received placebo orally for 10 weeks (period 1) followed by atorvastatin 20 mg orally for 10 weeks (period 2), separated by a 2-week washout period.
  Interventions: Drug: Atorvastatin; Drug: Placebo to Atorvastatin
- Part B: Ezetimibe (Active Comparator): Participants received 10 mg ezetimibe orally only a day and placebo to evolocumab by subcutaneous injection once a month for 24 weeks.
  Interventions: Drug: Ezetimibe; Other: Placebo to Evolocumab
- Part B: Evolocumab (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo to ezetimibe orally once a day for 24 weeks.
  Interventions: Other: Placebo to Ezetimibe; Drug: Evolocumab
- Part C: Open-label Evolocumab (Experimental): Participants who completed part B and were eligible to proceed to open-label extension part C and could choose quarterly between evolocumab 420 mg once a month or evolocumab 140 mg every 2 weeks for up to 2 years.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin was supplied as over-encapsulated 20 mg tablets
  Other Names: Lipitor
  Arms: Part A: Atorvastatin 20 mg => Placebo; Part A: Placebo => Atorvastatin 20 mg
Drug: Placebo to Atorvastatin — Placebo matching to atorvastatin supplied as over-encapsulated tablets
  Arms: Part A: Atorvastatin 20 mg => Placebo; Part A: Placebo => Atorvastatin 20 mg
Other: Placebo to Ezetimibe — Placebo matching to Ezetimibe supplied as over-encapsulated tablets.
  Arms: Part B: Evolocumab
Drug: Ezetimibe — Ezetimibe was supplied as 10 mg tablets, over-encapsulated for blinding.
  Other Names: Zetia
  Arms: Part B: Ezetimibe
Other: Placebo to Evolocumab — Placebo matching to evolocumab supplied as single-use prefilled autoinjector/pen(s)
  Arms: Part B: Ezetimibe
Drug: Evolocumab — Evolocumab supplied as single-use prefilled autoinjector/pen(s)
  Other Names: Repatha
  Arms: Part B: Evolocumab; Part C: Open-label Evolocumab

SUMMARY:
The primary objective of this study was to evaluate the effect of 24 weeks of evolocumab administered subcutaneously (SC) every month, compared with ezetimibe, on low-density lipoprotein cholesterol (LDL-C) levels in adults with high cholesterol who are unable to tolerate an effective dose of a statin due to muscle-related side effects (MRSE).

DETAILED DESCRIPTION:
The study is divided into 3 parts (A, B, C). After an initial 4-week washout period in which any statins, ezetimibe, or other lipid-lowering agents were discontinued, participants were enrolled in phase A, a double-blind, placebo-controlled crossover procedure to rechallenge patients with atorvastatin. Patients were randomly assigned in a 1:1 ratio to receive either atorvastatin (20 mg daily) or matching placebo for the first 10 weeks (period 1), then underwent a 2-week washout period, followed by crossover to the alternate therapy for a second 10-week period (period 2). Patients who experienced intolerable muscle symptoms during the first period did not complete the full 10 weeks of exposure but entered a 2-week washout period before proceeding to period 2.

Participants who did not develop muscle-related side effects were removed from the study, as were patients who reported muscle-related side effects during a placebo period.

After completion of phase A, patients who experienced muscle-related adverse effects while taking atorvastatin but not placebo were eligible for phase B, a 24-week, double-blind randomization to ezetimibe or evolocumab using a double-dummy design in which patients received either injectable placebo and oral ezetimibe or injectable evolocumab and oral placebo. A patient could proceed directly to phase B if they had a documented history of creatine kinase (CK) elevation more than 10 times the upper limit of normal accompanied by muscle symptoms while taking statin therapy, with documented resolution of both CK elevation and symptoms upon discontinuation of statin therapy.

These study procedures were designed to ensure that only patients with reproducible statin-associated muscle symptoms entered phase B of the study. For phase B, participants were randomized 2:1 to receive subcutaneously administered evolocumab (420 mg monthly) or oral ezetimibe (10 mg daily). Randomization in part B was stratified by screening LDL-C level (< 180 mg/dL [4.66 mmol/L] vs. ≥ 180 mg/dL) at study baseline.

Participants who completed phase B and did not discontinue SC investigational product for any reason, including an adverse event, were eligible to proceed to the 2-year open-label extension phase C to evaluate the long-term safety and efficacy of evolocumab in statin-intolerant patients. Participants in phase C were allowed to choose quarterly between evolocumab 420 mg SC QM or evolocumab 140 mg SC every 2 weeks (Q2W).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* Subject not at LDL-C goal
* History of statin intolerance
* Lipid lowering therapy has been stable prior to enrolment for at least 4 weeks
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes
* Poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (57):
- United States (18):
  - Research Site, Beverly Hills, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Pedro, California
  - Research Site, Atlanta, Georgia
  - Research Site, Sterling, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, York, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, Ashford, South Australia
- Canada (7):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- Czechia (2):
  - Research Site, Hradec Králové
  - Research Site, Prague
- Denmark (2):
  - Research Site, Aarhus N
  - Research Site, Glostrup Municipality
- France (3):
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Vénissieux
- Germany (3):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, München
- Italy (6):
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Cinisello Balsamo (MI)
  - Research Site, Ferrara
  - Research Site, Perugia
  - Research Site, Pisa
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
  - Research Site, Zwijndrecht
- Research Site, Christchurch, New Zealand
- Norway (2):
  - Research Site, Ålesund
  - Research Site, Oslo
- South Africa (4):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Midrand, Gauteng
  - Research Site, Observatory, Western Cape
  - Research Site, Parow, Western Cape
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Newcastle upon Tyne

REFERENCES:
- [Background] Cho L, Dent R, Stroes ESG, Stein EA, Sullivan D, Ruzza A, Flower A, Somaratne R, Rosenson RS. Persistent Safety and Efficacy of Evolocumab in Patients with Statin Intolerance: a Subset Analysis of the OSLER Open-Label Extension Studies. Cardiovasc Drugs Ther. 2018 Aug;32(4):365-372. doi: 10.1007/s10557-018-6817-7. PMID 30073585
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Nissen SE, Stroes E, Dent-Acosta RE, Rosenson RS, Lehman SJ, Sattar N, Preiss D, Bruckert E, Ceska R, Lepor N, Ballantyne CM, Gouni-Berthold I, Elliott M, Brennan DM, Wasserman SM, Somaratne R, Scott R, Stein EA; GAUSS-3 Investigators. Efficacy and Tolerability of Evolocumab vs Ezetimibe in Patients With Muscle-Related Statin Intolerance: The GAUSS-3 Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1580-90. doi: 10.1001/jama.2016.3608. PMID 27039291
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 511 participants were enrolled (492 in Part A and 19 directly in Part B) at 53 centers in the United States of America, Europe, Australia, New Zealand, Canada, and South Africa from December 2013 to November 2014.
  Results are reported for participants randomized in Part B. Part C was ongoing at the time of this analysis.
Pre-assignment Details: A total of 492 patients were randomized in part A; of those, 202 completed both periods and experienced muscle-related side effects during the atorvastatin period and not during the placebo period. Of the 202, 199 enrolled in Part B. Nineteen additional patients bypassed part A, as permitted by protocol, and advanced directly into part B.
Groups:
- Ezetimibe: Participants received 10 mg ezetimibe orally once a day and placebo to evolocumab by subcutaneous injection once a month for 24 weeks.
- Evolocumab: Participants received 420 mg evolocumab by subcutaneous injection once a month and placebo to ezetimibe orally once a day for 24 weeks.
Period: Overall Study
Arm/Group | Ezetimibe | Evolocumab
Started | 73 | 145
Completed | 70 | 138
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Evolocumab | Total
Number analyzed (Participants) | 73 | 145 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.4) | 59.0 (11.1) | 58.8 (10.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 52 | 92 | 144
  ≥ 65 years | 21 | 53 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 67 | 106
  Male | 34 | 78 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 73 | 143 | 216
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Black or African American | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 69 | 138 | 207
  Other | 0 | 2 | 2
Stratification Factor: Screening Low-density Lipoprotein Cholesterol (LDL-C) [Count of Participants; unit: Participants]
  < 180 mg/dL | 21 | 40 | 61
  ≥ 180 mg/dL | 52 | 105 | 157
LDL-C Concentation [Mean (Standard Deviation); unit: mg/dL] | 221.9 (70.2) | 218.8 (73.1) | 219.9 (72.0)
Total Cholesterol Concentration [Mean (Standard Deviation); unit: mg/dL] | 308.0 (73.8) | 306.5 (75.4) | 307.0 (74.7)
High-density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 50.2 (15.5) | 49.7 (15.4) | 49.8 (15.4)
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 35.7 (14.3) | 37.1 (15.6) | 36.7 (15.1)
Non-high-density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 257.8 (76.3) | 256.9 (73.8) | 257.2 (74.5)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 155.0 (42.4) | 158.3 (41.5) | 157.2 (41.7)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 6.709 (2.746) | 6.668 (2.349) | 6.682 (2.483)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] | 1.063 (0.416) | 1.063 (0.340) | 1.063 (0.366)
Triglyceride Concentration [Median (Inter-Quartile Range); unit: mg/dL] | 162.5 [127.0 to 231.0] | 176.0 [128.0 to 233.5] | 171.3 [127.0 to 233.0]
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L] | 38.0 [18.0 to 164.0] | 29.0 [12.5 to 152.5] | 31.0 [15.0 to 156.0]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -16.70 (1.91) | -54.50 (1.39)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; The null hypothesis was that there was no mean difference in the percent change from baseline at week 24 of part B or in the mean percent change from baseline at weeks 22 and 24 of part B in LDL-C between evolocumab 420 mg and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; p < 0.0001, Repeated Measures Model; Model includes treatment group, stratification factor (screening LDL-C), scheduled visit and interaction of treatment with scheduled visit; LS Mean Treatment Difference = -37.79, 95% CI 2-sided [-42.31 to -33.28], Standard Error of Mean 2.29

2. Primary Outcome: Percent Change From Baseline in LDL-C at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -16.69 (2.11) | -52.76 (1.52)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -36.07, 95% CI 2-sided [-41.07 to -31.08], Standard Error of Mean 2.53

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 22 and 24
Time Frame: Baselie and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
mg/dL | -31.0 (3.8) | -106.8 (2.7)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -75.8, 95% CI 2-sided [-84.7 to -67.0], Standard Error of Mean 4.5

4. Secondary Outcome: Change From Baseline in LDL-C at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
mg/dL | -31.2 (4.0) | -102.9 (2.9)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -71.7, 95% CI 2-sided [-81.3 to -62.2], Standard Error of Mean 4.8

5. Secondary Outcome: Percentage of Participants Who Achieved a Mean LDL-C at Weeks 22 and 24 of Less Than 70 mg/dL
Time Frame: Weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percentage of participants | 1.4 [0.3 to 7.7] | 29.9 [22.9 to 38.1]
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on Cochran-Mantel Haenszel test stratified by the stratification factor (screening LDL-C); Treatment Difference = 28.5, 95% CI 2-sided [19.1 to 36.7]

6. Secondary Outcome: Percentage of Participants Who Achieved LDL-C at Week 24 of Less Than 70 mg/dL
Time Frame: Week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percentage of participants | 0.0 [0.0 to 6.3] | 27.4 [20.1 to 36.1]
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on Cochran-Mantel Haenszel test stratified by the stratification factor (screening LDL-C); Treatment Difference = 27.4, 95% CI 2-sided [17.7 to 36.1]

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.43 (1.41) | -38.04 (1.03)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.61, 95% CI 2-sided [-29.95 to -23.27], Standard Error of Mean 1.69

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.57 (1.52) | -36.64 (1.10)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.08, 95% CI 2-sided [-28.67 to -21.48], Standard Error of Mean 1.82

9. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -14.38 (1.72) | -47.44 (1.25)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.06, 95% CI 2-sided [-37.12 to -28.99], Standard Error of Mean 2.06

10. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -14.62 (1.83) | -45.72 (1.32)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.10, 95% CI 2-sided [-35.44 to -16.76], Standard Error of Mean 2.20

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.42 (1.82) | -45.28 (1.31)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.86, 95% CI 2-sided [-38.15 to -29.58], Standard Error of Mean 2.17

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.74 (1.94) | -43.50 (1.40)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.75, 95% CI 2-sided [-36.35 to -27.16], Standard Error of Mean 2.33

13. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.48 (1.75) | -41.39 (1.27)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -29.91, 95% CI 2-sided [-34.06 to -25.77], Standard Error of Mean 2.10

14. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 173 | 145
percent change | -12.84 (1.85) | -40.04 (1.33)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.20, 95% CI 2-sided [-31.58 to -22.82], Standard Error of Mean 2.22

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at the Mean of Weeks 22 and 24
Time Frame: Baseline and Weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -11.86 (1.89) | -45.99 (1.36)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.13, 95% CI 2-sided [-38.59 to -29.67], Standard Error of Mean 2.26

16. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -12.62 (1.97) | -44.60 (1.41)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -31.98, 95% CI 2-sided [-36.64 to -27.32], Standard Error of Mean 2.36

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 22 and 24
Time Frame: Baseline and Weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -1.63 (2.80) | -22.71 (2.03)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.08, 95% CI 2-sided [-27.65 to -14.51], Standard Error of Mean 3.33

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | 0.17 (3.05) | -21.06 (2.19)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p < 0.0001, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.24, 95% CI 2-sided [-28.42 to -14.05], Standard Error of Mean 3.64

19. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -0.95 (3.94) | -5.39 (2.84)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.37, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -4.44, 95% CI 2-sided [-13.74 to 4.87], Standard Error of Mean 4.72

20. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -1.07 (4.97) | -2.88 (3.54)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.37, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.82, 95% CI 2-sided [-13.64 to 10.01], Standard Error of Mean 6.00

21. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at Week 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | 1.66 (1.71) | 7.85 (1.24)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.0083, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.18, 95% CI 2-sided [2.15 to 10.22], Standard Error of Mean 2.05

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | 2.90 (1.89) | 7.40 (1.36)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.0083, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 4.50, 95% CI 2-sided [0.02 to 8.98], Standard Error of Mean 2.27

23. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C) at the Mean of Weeks 22 and 24
Time Frame: Baseline and weeks 22 and 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -2.15 (3.22) | -6.81 (2.33)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.37, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -4.65, 95% CI 2-sided [-12.25 to 2.94], Standard Error of Mean 3.85

24. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 24
Time Frame: Baseline and week 24
Population: Participants randomized and dosed in Part B of the study
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab
Number analyzed (Participants) | 73 | 145
percent change | -2.66 (3.88) | -3.90 (2.78)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab; Test type: Superiority; p = 0.37, Repeated Measures Model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -1.23, 95% CI 2-sided [-10.45 to 7.98], Standard Error of Mean 4.67

ADVERSE EVENTS:
Time Frame: 6 months
Description: Results are reported for participants randomized in Part B. Adverse event data are not included for Part A as this phase was designed to ensure that only patients with reproducible statin-associated muscle symptoms entered Part B and was not the focus of the study. Part C was still ongoing at the time of this analysis.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Ezetimibe: Participants received 10 mg ezetimibe orally only a day and placebo to evolocumab by subcutaneous injection once a month for 24 weeks.
Arm/Group | Evolocumab | Ezetimibe
Serious Adverse Events (participants affected / at risk) | 9/145 | 10/73
Other Adverse Events (participants affected / at risk) | 80/145 | 40/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=145) | Ezetimibe (N=73)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Coronary artery perforation (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=145) | Ezetimibe (N=73)
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Fatigue (General disorders) | 12 | 5
Influenza like illness (General disorders) | 1 | 4
Bronchitis (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 14 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 1
Headache (Nervous system disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.